CLINICAL TRIAL: NCT05399134
Title: Glycemic Evaluation of Novel Staple Foods
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Responsible Party: Principal Investigator, Mei Hui Liu, Co-Investigator, National University of Singapore
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 2019/00952
Record Dates: First submitted 2022-05-23; First posted 2022-06-01 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2023-06

CONDITIONS: Diabete Type 2; Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: A within-subject crossover study design is used to assess the effectiveness of incorporating novel staple food into people's diet to improve their glycemic control. Subjects will undergo two study arms: Treatment and Control. The duration of each arm is 14-days, with a 1-week washout period in between.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Modified Functional Foods (Treatment) (Experimental): Anthocyanin black rice extract powder (ABREP)-fortified bread, microfluidic co-flow noodles, and 5ibrePlus™-fortified white rice for breakfast, lunch, and dinner respectively served in a mixed meal.
  Interventions: Dietary Supplement: Modified Functional Foods
- Control Functional Foods (Control) (Placebo Comparator): White bread, beehoon noodles, and jasmine white rice for breakfast, lunch, and dinner respectively served in a mixed meal.
  Interventions: Dietary Supplement: Control Functional Foods

INTERVENTIONS:
Dietary Supplement: Modified Functional Foods — Subjects will be provided with ABREP-fortified bread, microfluidic co-flow noodles, and 5ibrePlus™-fortified white rice served in a mixed meal.
  ABREP-fortified bread: Anthocyanins are known to exert anti-diabetic effects through modulating digestion, glucose uptake, insulin secretion and sensitivity. Moreover, inhibitory effects of anthocyanins on various carbohydrases, including a-glucosidase and a-amylase have been widely reported.
  Microfluidic co-flow noodles: Microfluidic technology is employed to design noodle-food structures consisting of a mix of soy protein isolate and alginate as gelling agents to offer a type of novel noodles with proteins and negligible carbohydrate content.
  5ibrePlus™-fortified white rice: 5ibrePlus™ is a patented novel fibre grain product by Alchemy Foodtech Pte. Ltd (WO 2017/142477) with reduced GI. Its main constituents are insoluble resistant starch and soluble fibre.
  Arms: Modified Functional Foods (Treatment)
Dietary Supplement: Control Functional Foods — Subjects will be provided with control function foods including white bread, beehoon noodles, and jasmine white rice served in a mixed meal.
  Arms: Control Functional Foods (Control)

SUMMARY:
In this study, the combined effects of functional foods (i.e. Anthocyanin fortified bread, Microfluidic co-flow noodles, 5ibrePlus™-fortified white rice) is investigated in an ad-libitum diet and their contributions to diabetes management.

DETAILED DESCRIPTION:
Research has confirmed that a food's glycemic effect cannot be accurately predicted from the type and amount of carbohydrates it contains, as the rate at which the carbohydrates is digested and released into the bloodstream is influenced by many factors such as the food's physical form, its fat, protein and fibre content, and the chemical structure of its carbohydrates. For these reasons, it is possible to produce food from the same group with different effects on blood glucose. Consumption of low GI food has shown to improve glycemic control, lipid profile and reduce systemic inflammation. With bread, noodles and rice being the staple food for many Singaporeans, functional staple food alternatives offer a lower GI alternative without greatly affecting the population's dietary preference. Preliminary studies for each functional staple food alternative (for bread, noodles, and rice) had reflected improved glycaemic responses compared to their staple counterparts.

ELIGIBILITY:
Inclusion Criteria:

* Chinese ethnicity
* English-speaking
* Age between 21 - 70 years old inclusive.
* Confirmed Type 2 Diabetes with HbA1c level of less than 10%
* Not on prandial insulin therapy
* Subjects with stable medical problems not limited to hypertension and hyperlipidemia

Exclusion Criteria:

* Current smoker or use of tobacco products within the 3 months
* Vegetarian or other dietary restrictions that would not allow the subject to consume the test meal.
* Persons with electronic medical implants (e.g. pacemaker).
* Persons with known or ongoing psychiatric disorders or drug abuse within 3 years.
* Women who are pregnant or lactating.
* Persons with an average weekly alcohol intake that exceeds 21 units per week (males) and 14 units per week (females). 1 unit is equivalent to:

  * 12 oz or 360 mL of beer;
  * 5 oz or 150 mL of wine;
  * 1.5 oz or 45 mL of distilled spirits.
* Persons with active infection(s) requiring systemic, antiviral or antimicrobial therapy that will not be completed prior to the first study visit
* Persons who have undergone treatment with any investigational drug or biological agent within one (1) month of screening or plans to enroll in another study involving investigational drugs/biological agents during the duration of this study.
* Persons with significant change in weight (+/- 5%) during the past month.
* Persons with a known allergy to rice bran, dietary fiber, alginate and other study components (anthocyanins, soy protein).

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-05-19 (Actual); Study Completion 2023-05-19 (Actual)

PRIMARY OUTCOMES:
Postprandial glycemic response of novel staple foods in Type 2 diabetics | 5 weeks
  Incremental area under the curve (iAUC) post prandial glycemic response from continuous glucose monitoring of diet incorporated with novel staple foods, in comparison to control staple foods, in Type 2 diabetic individuals.

CONTACTS AND LOCATIONS:
Overall Officials: Mei Hui Liu, Principal Investigator — National University of Singapore
Locations (1):
- National University of Singapore, Singapore, Singapore, Singapore